CLINICAL TRIAL: NCT07229482
Title: Cardiometabolic Effects of a Potato-rich Diet in Older Adults at Increased Risk of Developing Type 2 Diabetes: A Randomized Controlled Feeding Study
Brief Title: Potatoes, Type 2 Diabetes, and Cardiometabolic Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Dennis Cladis, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25-897
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: T2D; Blood Pressure; Cardiometabolic Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato-rich healthy diet pattern (Experimental): Following a 2-week eucaloric lead-in diet, participants will be provided and consume a potato-rich healthy dietary pattern for 12 weeks.
  Interventions: Other: Controlled diet: Potato-rich healthy dietary pattern
- Typical Western-style dietary pattern (Active Comparator): Following a 2-week eucaloric lead-in diet, participants will be provided and consume a typical Western-style dietary pattern for 12 weeks.
  Interventions: Other: Controlled diet: Typical Western-style dietary pattern

INTERVENTIONS:
Other: Controlled diet: Potato-rich healthy dietary pattern — Following a 2-week eucaloric lead-in diet, participants will be provided and consume a potato-rich healthy dietary pattern for 12 weeks. The intervention diet will be eucaloric and matched for macronutrient composition with the control diet. Whole white potatoes will be incorporated into the intervention diet in different forms. This diet will have an healthy eating index (HEI) score of 85.
  Arms: Potato-rich healthy diet pattern
Other: Controlled diet: Typical Western-style dietary pattern — Following a 2-week eucaloric lead-in diet, participants will be provided and consume a typical Western-style dietary pattern for 12 weeks. The control diet will be potato-free, eucaloric, and matched for macronutrient composition with the intervention diet. This diet will have an healthy eating index (HEI) score of 58.
  Arms: Typical Western-style dietary pattern

SUMMARY:
Type 2 diabetes (T2D) is a major chronic health condition which increases risk of coronary artery disease, frailty, cognitive decline, and mortality. Additionally, hypertension is a major comorbidity for individuals with T2D, further increasing the risk of adverse cardiovascular outcomes. The prevalence of both conditions increases with advancing age. There is an urgent need to identify new approaches to prevent the development of T2D and improve cardiometabolic health in older adults 50-70 years of age.

Whole white potatoes are an unprocessed food rich in essential nutrients often under-consumed by Americans, including potassium, fiber, magnesium, vitamins C and B6, and phytochemicals. Each of these nutrients individually are associated with cardiometabolic health benefits. Potatoes account for a significant amount of the intake of these nutrients in the US diet and are well-positioned to be a foundational element of a healthy dietary pattern. However, there are few interventional studies evaluating the effect of potatoes on cardiometabolic health, and the evidence from observational studies is mixed, leaving a significant gap in knowledge regarding the potential for potatoes to be included in healthy dietary patterns.

The results of our proposed study will provide foundational data that inform future dietary guidelines regarding the inclusion of white potatoes as part of a healthy US dietary pattern.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-70 years
* Weight stable for previous 3 months (±5% body weight)
* Sedentary to recreationally active
* ADA-Risk Screener questionnaire score of at least 5
* No plans to gain or lose weight or change physical activity level
* Willing to pick up food daily and consume foods provided for a 14-week period
* Verbal and written informed consent
* Estrogen or testosterone use, lipid-lowering medication and thyroid replacement medication is acceptable, if on stable dose for >6 months

Exclusion Criteria:

* Body mass index >40 m2/kg
* Diabetes or diabetes medication
* Weight loss medication or medication influencing glucose metabolism
* Antibiotic, prebiotic or probiotic use in prior 3 months
* TCHOL >6.2 mmol/L; TG >4.5 mmol/L
* Blood pressure (BP) > 159/99 mmHg or taking antihypertensive medication
* Diagnosed inflammatory bowel disease
* Past or current heart diseases, stroke, respiratory disease, endocrine or metabolic disease, or hematological-oncological disease
* Vegetarian or vegan
* Pregnant or plans to become pregnant
* Food allergies or aversions to diet foods provided
* Estrogen or testosterone usage or lipid-lowering medication usage <6 months

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in glucose tolerance from baseline to 12 weeks post potato-rich healthy diet vs typical Western-style diet | 2-hour test in laboratory, 2 timepoints (baseline, 12-weeks post intervention diets)
  Glucose tolerance will be assessed using a 2-hour oral glucose tolerance test (OGTT, 75 g glucose load). Blood will be collected at baseline (fasting) and thereafter at 30-minute intervals (5 total measurements in 2 hours).
Change in insulin sensitivity from baseline to 12 weeks post potato-rich healthy diet vs typical Western-style diet | 2-hour test in laboratory, 2 timepoints (baseline, 12-weeks post intervention diets)
  Insulin sensitivity will be assessed using a 2-hour oral glucose tolerance test (OGTT, 75 g glucose load). Blood will be collected at baseline (fasting) and thereafter at 30-minute intervals (5 total measurements in 2 hours).
Change in glucose control (AUC) from baseline to 12 weeks post potato-rich healthy diet vs typical Western-style diet | 7-day measurement during free-living, 2 timepoints (baseline, 12 weeks post intervention diets)
  24-hour glucose control (24-hour AUC) will be assessed using continuous glucose monitoring for a 7-day period.
Change in blood pressure from baseline to 12 weeks post potato-rich healthy diet vs typical Western-style diet | 20-minute measurement in the laboratory, 2 timepoints (baseline, post 12 week intervention diets)
  Seated, resting blood pressure will be measured via automated sphygmomanometry, according to American Heart Association guidelines. Both diastolic and systolic blood pressures will be measured.

SECONDARY OUTCOMES:
Change in inflammatory biomarker tumor necrosis factor alpha from baseline to 12 weeks post potato-rich healthy diet vs typical Western-style diet | 5-minute blood collection in laboratory, 2 timepoints (baseline, post 12 week intervention diets)
  Tumor necrosis factor alpha will be measured in fasting blood samples via ELISA kits.
Change in inflammatory biomarker interleukin-6 from baseline to 12 weeks post potato-rich healthy diet vs typical Western-style diet | 5-minute blood collection in laboratory, 2 timepoints (baseline, post 12 week intervention diets)
  Inflammatory biomarker interleukin-6 will be measured in fasting blood samples via ELISA kits.
Change in inflammatory biomarker monocyte chemoattractant protein-1 from baseline to 12 weeks post potato-rich healthy diet vs typical Western-style diet | 5-minute blood collection in laboratory, 2 timepoints (baseline, post 12 week intervention diets)
  Inflammatory biomarker monocyte chemoattractant protein-1 will be measured in fasting blood samples via ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Cladis, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Polytechnic Institute and State University, Blacksburg, Virginia, United States